CLINICAL TRIAL: NCT05947071
Title: Comparison of High vs Standard Dose Influenza Vaccines in Pediatric Solid Organ Transplant Recipients
Brief Title: High vs.Standard Dose Influenza Vaccine in Pediatric Solid Organ Transplant (SOT) Recipients
Acronym: PSOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DAIT RTB-019
Record Dates: First submitted 2023-03-01; First posted 2023-07-17 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Immunization; Infection; Transplantation Infection; Influenza
Keywords: Influenza; Vaccination; Immunization; High Dose; Fluzone; Standard Dose; Influenza, Human; Communicable Diseases; Pediatric transplantation
MeSH Terms: conditions — Infections; Influenza, Human; Communicable Diseases | interventions — Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Intervention Model Description: The primary goal of this two-arm, double blind, randomized controlled trial is to compare influenza vaccine immunogenicity and safety between (a) two doses of SD-QIV and (b) two doses of HD-QIV over one influenza season in a population of pediatric SOT recipients who are ≥1 month and <24 months post-transplant at the time of study immunization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study staff, and subjects will be blinded to which vaccine the subject will receive, except for an un-blinded vaccinator. This individual will not inform the study team or the subjects which vaccine they administered to the subject. The un-blinded vaccinator will not participate in any other study activities. The pharmacy will be un-blinded and will have a record of which vaccine was given to each subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Two Doses Standard Dose Quadrivalent Inactivated Influenza Vaccine (Experimental): Two doses of SD-QIV (0.5 mL; 15µg of each influenza antigen) 28-42 days apart
  Interventions: Biological: Standard Dose Quadrivalent Inactivated Influenza Vaccine
- Two Doses High Dose Quadrivalent Inactivated Influenza Vaccine (Experimental): Two doses of HD-QIV (0.7 mL; 60µg of each influenza antigen) 28-42 days apart
  Interventions: Biological: High Dose Quadrivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Standard Dose Quadrivalent Inactivated Influenza Vaccine — Fluzone ® Quadrivalent is a vaccine indicated for active immunization for the prevention of influenza disease caused by two influenza A subtype viruses and two type B viruses contained in the vaccine.
  Other Names: Fluzone
  Arms: Two Doses Standard Dose Quadrivalent Inactivated Influenza Vaccine
Biological: High Dose Quadrivalent Inactivated Influenza Vaccine — Fluzone High-Dose (Influenza Vaccine) for intramuscular injection is an inactivated influenza vaccine, prepared from influenza viruses propagated in embryonated chicken eggs. The virus-containing allantoic fluid is harvested and inactivated with formaldehyde. Influenza virus is concentrated and purified in a linear sucrose density gradient solution using a continuous flow centrifuge. The virus is then chemically disrupted using a non-ionic surfactant, octylphenol ethoxylate (Triton® X-100), producing a "split virus". The split virus is further purified and then suspended in sodium phosphatebuffered isotonic sodium chloride solution. The Fluzone High-Dose process uses an additional concentration factor after the ultrafiltration step in order to obtain a higher hemagglutinin (HA) antigen concentration.
  Other Names: Fluzone High Dose
  Arms: Two Doses High Dose Quadrivalent Inactivated Influenza Vaccine

SUMMARY:
Influenza virus is a significant pathogen in pediatric solid organ transplant (SOT) recipients. However, these individuals respond poorly to standard-dose (SD) inactivated influenza vaccine (IIV). Recent studies have investigated two strategies to overcome poor immune responses in SOT recipients: (1) administration of high-dose (HD)-IIV compared to SD-IIV and (2) two doses of SD-IIV compared to one dose of SD-IIV in the same influenza season. One study compared HD-IIV vs. SD-IIV in adult SOT recipients and noted that HD-IIV was safe and more immunogenic; however, the median post-transplant period was 38 months. A phase I pediatric study comparing a single dose of HD-IIV vs. SD-IIV was safe with higher immunogenicity, but the study was limited by small sample size and median post-transplant vaccine administration was 26 months. In another phase II trial of adult SOT recipients, two doses of SD-IIV one month apart compared to one-dose of SD-IIV revealed modestly increased immunogenicity when given at a median of 18 months post-transplant. Therefore, these studies lack both evaluation in the early post-transplant period and substantive pediatric populations. Additionally, the administration of two-doses of HD-IIV in the same influenza season has not been evaluated in pediatric SOT recipients. Thus, the optimal immunization strategy for pediatric SOT recipients less than 24 months post-transplant is unknown. In addition, immunologic predictors and correlates of influenza vaccine immunogenicity in pediatric SOT recipients have not been well-defined.

The central hypothesis of our proposal is that pediatric SOT recipients 1-23 months post-transplant who receive two doses of HD-quadrivalent inactivated influenza vaccine (QIV) will have similar safety but higher Hemagglutination Inhibition (HAI) geometric mean titers (GMTs) to influenza antigens compared to pediatric SOT recipients receiving two doses of SD-QIV.

DETAILED DESCRIPTION:
Study design: This is a phase II, multi-center, double-blind, randomized controlled immunogenicity and safety trial comparing two doses of HD-QIV or two doses of SD-QIV in pediatric SOT recipients.

Hypotheses:

1. Pediatric SOT recipients who are 1-23 months out from transplant and are administered two doses of HD-QIV will develop higher Hemagglutination Inhibition (HAI) geometric mean titer (GMT) to influenza antigens compared to pediatric SOT recipients receiving two doses of SD-QIV, with Geometric Mean Titer Ratio (GMR) HD-QIV/SD-QIV greater than 1.0.
2. Administration of HD-QIV in pediatric SOT recipients will be well tolerated and the safety profile will be similar to SD-QIV with regards to solicited local and systemic post-administration reactions.
3. Baseline immunophenotypic markers of exhaustion, immune senescence, and immune activation at the pre-vaccine timepoint will correlate with post-vaccine HAI titers.

Study population: The study plans to enroll a total of approximately 312 pediatric heart, liver, and/or kidney transplant recipients between 1 and 23 months post-transplantation.

Study enrollment: The enrollment period will be over three-years. Participants will be randomized into one of two groups. Group 1 will receive two doses of SD-QIV (0.5 mL; 15μg of each influenza antigen) whereas Group 2 will receive two doses HD-QIV (0.7 mL; 60μg of each influenza antigen).

Influenza surveillance: Active surveillance for influenza-like symptoms will begin when influenza season starts in each site's community, defined in previous trials as identification of at least two positive respiratory tests for influenza, with at least 10% of diagnostic tests positive during two consecutive weeks in the local clinical or research laboratory. Enrollment will continue during influenza season with nasal swabs obtained at all main visits to document the occurrence of influenza virus both prior to and after vaccination. During the influenza season, the study staff will attempt to do a weekly telephone and/or electronic communication with the participants to detect and document any influenza-like illness (ILI) and any specific coronavirus disease of 2019 (COVID-19) like symptoms.

If participants meet ILI criteria and/or any specific coronavirus disease of 2019 (COVID-19) like symptoms (see below), an additional nasal swab will be collected*.

ILI criteria are met by occurrence of one of the conditions below:

* Fever: ≥38°C (100.4°F)
* Two or more of any of the following: respiratory symptoms (rhinorrhea, sinus congestion, post-nasal drip, shortness of breath, cough, wheezing, sputum production, sore throat, sneezing, watery eyes, ear pain, hoarseness); or systemic symptoms (myalgias, chills, chest pain, or headache); or new loss of taste or new loss of smell; or gastrointestinal symptoms (diarrhea or vomiting).

  * Per investigators' discretion at each individual site, a swab is not needed if there is a known non-respiratory cause of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 3-17 years of age at time of enrollment
2. Pediatric kidney, heart, and/or liver transplant recipient ≥1 month and <24 months post-transplant at the time of study immunization

   * Note: Inclusion of recipients of multiple organs is permitted but is limited to recipients of any combination of organs including kidney, heart and/or liver
   * Note: Participants undergoing re-transplantation are permitted
3. Anticipated to be available for duration of the study
4. Available by telephone, email, or text message

Exclusion Criteria:

1. Inability (i.e. not able to understand and provide consent) or unwillingness of a participant/parent/legal guardian to give written informed consent or comply with study protocol
2. History of severe hypersensitivity to influenza vaccination or anaphylaxis to eggs/egg protein
3. History of severe latex hypersensitivity
4. History of Guillain-Barre syndrome
5. History of lung or intestine transplant
6. HIV positive patients (testing within 24 months of enrollment)
7. Receipt of current season's influenza vaccine post-transplant prior to enrollment in the study
8. Currently pregnant or lactating (females of childbearing age may be enrolled based on self-report, urine pregnancy test must be performed prior to each influenza vaccine)
9. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity: Hemagglutination Inhibition (HAI) titers | 4 weeks following the 2nd study vaccine
  Antibody titers will be measured by hemagglutination inhibition assay.
Safety: solicited local and systemic post-administration reactions | in the first 7 days following each study vaccine
  Post-vaccination local adverse events (pain, tenderness, swelling/induration, erythema/redness, swelling/induration size, and erythema/redness size) and systemic adverse events (Fatigue/malaise, headache, nausea, body ache/myalgia (not at the injection site), general activity level, vomiting, and fever).

SECONDARY OUTCOMES:
Immunogenicity: Hemagglutination Inhibition (HAI) titers | 4 weeks following 1st and 2nd doses of each study vaccine
  Antibody titers will be measured by hemagglutination inhibition assay.
The number of participants achieving seroprotection and seroconversion for influenza virus. | 4 weeks following the 1st and 2nd study vaccination
  Antibody titers will be measured by hemagglutination inhibition assay. Seroconversion is defined as ≥ 4-fold rise in hemagglutination inhibition assay titers. Seroprotection is defined as ≥1:40 hemagglutination inhibition assay titer.
Durability of immunogenicity | 180 days after vaccine 2
  Measured as Hemagglutination Inhibition (HAI) titer at end of season

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Stanford University, Stanford, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No